CLINICAL TRIAL: NCT03364556
Title: Nutritional Intake and Bone Health Among Adults With Undiagnosed, Untreated Celiac Disease
Brief Title: Nutritional Intake and Bone Health in Celiac Disease
Status: Completed | Type: Observational
Sponsor: George Mason University (Other)
Responsible Party: Sponsor
Other Study IDs: 1159415
Record Dates: First submitted 2017-11-27; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention

SUMMARY:
Celiac disease leads to malnutrition and secondary conditions including osteoporosis. The dietary habits of adults with untreated, undiagnosed celiac disease has not yet been observed, but presents a critical piece in understanding the effects of the disease on bone health. Objective was to evaluate differences in nutritional intake of calcium, vitamin D, and phosphorus; serologic indices of these nutrients; and bone health among adults with and without celiac disease. Cross-sectional data from What We Eat in America (WWEIA) and the National Health and Nutrition Examination Survey (NHANES) 2009-14 was analyzed.

DETAILED DESCRIPTION:
Celiac disease leads to malnutrition and secondary conditions including osteoporosis. The dietary habits of adults with untreated, undiagnosed celiac disease has not yet been observed, but presents a critical piece in understanding the effects of the disease on bone health. Objective was to evaluate differences in nutritional intake of calcium, vitamin D, and phosphorus; serologic indices of these nutrients; and bone health among adults with and without celiac disease.

Cross-sectional data from What We Eat in America (WWEIA) and the National Health and Nutrition Examination Survey (NHANES) 2009-14 was analyzed, including self-reported dietary and supplement intake from one day of 24-hour recalls, serologic indicators, and dual x-ray absorptiometry (DXA) scans were analyzed in adults (n=49) testing positive for celiac disease to the tissue transglutaminase endomysial antibody assay (tTG-EMA). Statistical analysis included multiple linear regression modelling controlled for age, sex, race/ethnicity, energy intake, and poverty income ratio.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18+ years with a complete 24-hour recall in WWEIA and a completed celiac disease serologic test. Two groups were used in the analysis. The control group consisted of a normal adult population without celiac disease, as indicated by a negative serologic test for celiac disease and no self-reported celiac disease. The serologically positive group were considered to have undiagnosed, untreated celiac disease based on a positive serologic test for celiac disease (EMA+), no self-reported celiac disease, and no adherence to a gluten-free diet. NHANES employs two steps of serologic tests for selected participants to screen for celiac disease antibodies that develop as a T-cell-mediated response to gluten.

Exclusion Criteria:

* Adults were excluded if they were pregnant or breastfeeding at the time of the study, or if they reported any history of celiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18+ years with a complete 24-hour recall in WWEIA and a completed celiac disease serologic test. Two groups were used in the analysis. The control group consisted of a normal adult population without celiac disease, as indicated by a negative serologic test for celiac disease and no self-reported celiac disease. The serologically positive group were considered to have undiagnosed, untreated celiac disease based on a positive serologic test for celiac disease (EMA+), no self-reported celiac disease, and no adherence to a gluten-free diet. NHANES employs two steps of serologic tests for selected participants to screen for celiac disease antibodies that develop as a T-cell-mediated response to gluten.
Sampling Method: Probability Sample
Enrollment: 13893 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Dietary Intake | 24 hours
  24 hour recall

SECONDARY OUTCOMES:
Bone Mineral Density | Baseline
  DXA

IPD SHARING:
Plan to Share IPD: No
NHANES is publicly available data. No data sharing plan is needed.